CLINICAL TRIAL: NCT03879239
Title: A Prospective, Randomized, Multi-center, Double-Blinded, Placebo-Controlled, 3-Arm Clinical Study to Assess the Efficacy and Safety of Vibrant Capsule, for the Treatment of Chronic Idiopathic Constipation
Brief Title: Efficacy and Safety of Vibrant Capsule vs. Placebo for the Treatment of Chronic Idiopathic Constipation
Acronym: Vibrant
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vibrant Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 270CLD
Record Dates: First submitted 2019-02-17; First posted 2019-03-18 (Actual); Results first posted 2024-08-09 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Chronic Idiopathic Constipation

STUDY DESIGN:
Intervention Model Description: The study design initially comprised 3 arms: 2 active vibrating capsule arms (Modes A and B) and 1 placebo arm. Based on the analysis of the first pre-define phase of the study, active mode B was discontinued and the trial was completed using mode A. Therefore, study results are available only for active A and Placebo arms.
Who Masked: Participant, Investigator
Masking Description: This was a double blind, placebo controlled study and both the participant and the investigator were masked. The study investigators, sponsors and participants were all blinded throughout the study. A research pharmacist/investigator who was not involved with evaluating patients or conducting the study, provided training to the participants and dispensed the correct study arm allocation. This individual had no other role in the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (3):
- Vibrant Capsule mode A (Active Comparator): Vibrant Capsule mode A administered 5 times per week
  Interventions: Device: Vibrating capsule
- Vibrant Capsule mode B (Active Comparator): Vibrant Capsule mode B administered 5 times per week.
  Based on the analysis of the first pre-define phase of the study, active mode B was discontinued, and the trial was completed using mode A. Therefore, study results are not available for arm B.
  Interventions: Device: Vibrating capsule
- Placebo Capsule (Placebo Comparator): Placebo Capsule administered 5 times per week
  Interventions: Device: Vibrating capsule

INTERVENTIONS:
Device: Vibrating capsule — Vibrating Capsule administered 5 times per week

SUMMARY:
The study is a prospective, randomized, multicenter, adaptive design, double blinded, placebo-controlled study, to evaluate the efficacy and safety of Vibrant Capsule vs. placebo in relieving constipation in subjects with Chronic Idiopathic Constipation.

DETAILED DESCRIPTION:
Subjects came for 4 visits: Screening (visit 1), baseline (visit 2), after 4 treatment weeks from baseline (visit 3) and after 8 treatment weeks from baseline (Final visit , visit 4). A total of 8 treatment weeks

Three arms were assessed:

* Vibrant Capsule mode A administered 5 times per week
* Vibrant Capsule mode B administered 5 times per week
* Placebo Capsule administered 5 times per week The difference between the 2 operating modes is in the vibrating sequence during the capsule's operating time.

Following Interim Analysis one active arm was dropped and the study continued with 2 arms, placebo and an active arm.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects aged 22 years and older
2. Subjects with Chronic Idiopathic Constipation (CIC) according to Rome III criteria and who have not experienced relief of their symptoms from available therapies (osmotic and stimulant laxatives used for at least one month at recommended dose)
3. Subjects with an average of ≤2.5 Spontaneous Bowel Movements (SBM) per week and ≥1 SBM per week
4. Normal colonoscopy performed within 5 years prior to study participation, unless the subjects are <50 years old and without alarm signs and/or symptoms
5. Subject signed the Informed Consent Form (ICF)
6. Female subjects must have a negative blood pregnancy test during screening, confirmed by a negative urine pregnancy test during baseline and must not be lactating prior to receiving study medication. For females of child-bearing potential, a hormonal (i.e., oral, implantable, or injectable) and single-barrier method, or a double-barrier method of birth control must be used throughout the study. All other female subjects must have the reason for their inability to bear children documented in the medical record [i.e., tubal ligation, hysterectomy, or post-menopausal (defined as a minimum of one year since the last menstrual period)]; in these circumstances, a pregnancy test will not be necessary

Exclusion Criteria:

History of complicated/obstructive diverticular disease 2. History of intestinal or colonic obstruction, or suspected intestinal obstruction.

3. History of significant gastrointestinal disorder, including any form of inflammatory bowel disease or gastrointestinal malignancy (celiac disease is accepted if the subject has been treated and is in remission) 4. History of gastroparesis 5. Use of any of the following medications:

* Medications that may affect intestinal motility, prokinetics, anti-Parkinsonian medications, opiates, opioids, calcium-channel blockers, aluminum/magnesium hydroxide
* With the exception of antidepressants, thyroid or hormonal replacement therapy, when the subject has been on a stable dose for at least 3 months prior to enrollment.

  6. Clinical evidence of significant respiratory, cardiovascular, renal, hepatic, biliary, endocrine, psychiatric or neurologic disease 7. Presence of cardiac pacemaker or gastric electrical stimulator. 8. History of, or current eating disorders, such as anorexia, bulimia, or compulsory overeating.

  9. Diagnosis of mega-rectum or colon, congenital anorectal malformation, clinically significant rectocele, history of intestinal resection (with an exception for appendectomy, cholecystectomy and inguinal hernia repair), history of bariatric surgery or evidence of any structural abnormality of the gastrointestinal tract that might affect transit 10. History of Zenker's diverticulum, dysphagia, Barrett's esophagus, esophageal stricture or achalasia 11. Chronic use of non-steroidal anti-inflammatory drugs (NSAIDs): chronic use is defined as taking full dose NSAIDs more than three times a week for at least six months. Subjects on cardiac doses of aspirin may be enrolled in the study 12. Subjects with pelvic floor dysfunction/defecatory disorder, based on subject history 13. Participation in another clinical study within one month prior to screening.

  14. Women who are pregnant or lactating 15. Use of any medication for constipation relief during the study, except as rescue medication, as indicated by study rules 16. Inability to use an electronic daily Diary (on a computer, phone application, tablet or other electronic device) to report bowel movements, symptoms and medication usage 17. Subject participated in a previous Vibrant study 18. Subjects planning to undergo MRI during the study 19. Any known allergy to soybean or beeswax or Calcium Carbonate 20. Any other condition which in the opinion of the investigator may adversely affect the safety of the subject or would limit the subject's ability to complete the study

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 349 (Actual)
Dates: Start 2019-04-08 (Actual); Primary Completion 2021-07-16 (Actual); Study Completion 2022-01-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tal Malina, MBA, Study Director — Vibrant Ltd.
Locations (8):
- United States (8):
  - G & L Research, LLC., Foley, Alabama
  - Del Sol Research Management, Tucson, Arizona
  - Augusta University, Augusta, Georgia
  - PharmQuest, Greensboro, North Carolina
  - Great Lakes Medical Research LLC, Beachwood, Ohio
  - Clinical Inquest Center Ltd, Huber Heights, Ohio
  - Great Lakes Gastroenterology Research, Mentor, Ohio
  - Clinical Neuroscience Solutions dba CNS Healthcare, Memphis, Tennessee

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rao SSC, Quigley EMM, Chey WD, Sharma A, Lembo AJ. Randomized Placebo-Controlled Phase 3 Trial of Vibrating Capsule for Chronic Constipation. Gastroenterology. 2023 Jun;164(7):1202-1210.e6. doi: 10.1053/j.gastro.2023.02.013. Epub 2023 Feb 21. PMID 36822371
- [Derived] Rao SSC, Lembo A, Chey WD, Friedenberg K, Quigley EMM. Effects of the vibrating capsule on colonic circadian rhythm and bowel symptoms in chronic idiopathic constipation. Neurogastroenterol Motil. 2020 Nov;32(11):e13890. doi: 10.1111/nmo.13890. Epub 2020 May 25. PMID 32449277

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 95 centers in the USA. Recruitment began on 8 Apr 2019 and concluded on 16 July 2021.
Pre-assignment Details: Following the consent process, subjects who met the study criteria started a run-in period of 2-4 weeks, during which they completed a daily eDiary with questions regrading their bowel movements and constipation symptoms.
Groups:
- Vibrant Capsule Mode B: Vibrant Capsule mode B administered 5 times per week
  Vibrating capsule: Vibrating Capsule administered 5 times per week
Period: Overall Study
Arm/Group | Vibrant Capsule Mode A | Vibrant Capsule Mode B | Placebo Capsule
Started | 163 | 37 | 149
Completed | 141 | 30 | 133
Not Completed | 22 | 7 | 16

BASELINE CHARACTERISTICS:
Groups:
- Vibrant Capsule Mode B: Vibrant Capsule mode B administered 5 times per week. Based on the analysis of the first pre-define phase of the study Arm B was discontinued.
- Total: Total of all reporting groups
Arm/Group | Vibrant Capsule Mode A | Vibrant Capsule Mode B | Placebo Capsule | Total
Number analyzed (Participants) | 163 | 37 | 149 | 349
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.1 (13.33) | 45 (12.25) | 45.9 (13.47) | 46.4 (13.26)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 143 | 28 | 126 | 297
  Male | 20 | 9 | 23 | 52
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 77 | 22 | 60 | 159
  Hispanic or Latino | 31 | 3 | 34 | 68
  Black or African American | 41 | 11 | 39 | 91
  Asian/ Pacific Islander | 10 | 1 | 12 | 23
  Other | 4 | 0 | 4 | 8
Duration of constipation (years) [Mean (Standard Deviation); unit: years] — History of Constipation: presents the history of constipation parameters for all the subjects enrolled (3 study arms).
  years | 17.90 (14.15) | 11.20 (10.00) | 14.50 (12.35) | 15.80 (13.17)

OUTCOME MEASURES:

1. Primary Outcome: CSBM1 & CSBM2 Success Rate
Description: CSBM1Success Rate: defined as the number of subjects with an increase from the run-in period of at least one weekly Complete Spontaneous Bowel Movement (CSBM) during at least 6 of the 8 weeks of treatment.
  CSBM2 success rate: defined as the number of subject with an increase from the run-in period of at least two weekly Complete Spontaneous Bowel Movement (CSBM) during at least 6 of the 8 weeks of treatment.
  The study will be deemed successful if either the CSBM1 or the CSBM2 success rate is statistically significantly higher in the active arm that was continued after the interim analysis (Vibrant Capsule Mode A), than in the placebo arm
  NOTE:
  * A spontaneous bowel movement (SBM) is defined as a bowel movement that occurs at least 48h after laxative/rescue intake and without digital maneuver.
  * A complete spontaneous bowel movement (CSBM) is defined as a spontaneous bowel movement associated with a feeling of complete evacuation by the subject.
Time Frame: 8 weeks of treatment
Population: A predefined first-phase analysis was included in the protocol and approved by the FDA. The objective of this first phase analysis was to identify which of the 2 activation modes was superior, and to recommend that mode for the remainder of the study.
  Based on the analysis of the study's first phase, mode B was discontinued, and the trial was completed using mode A.
  Hence, per the pre-specified outcomes definition, the results are available for mode A &Placebo arms without the dropped Arm B.
Measure: Count of Participants; unit: Participants
Arm/Group | Vibrant Capsule Mode A | Placebo Capsule
Number analyzed (Participants) | 163 | 149
Participants
  CSBM1 Success Rate | 64 | 33
  CSBM2 Success Rate | 37 | 17
Statistical Analysis 1: Comparison: Vibrant Capsule Mode A vs Placebo Capsule; Test type: Superiority; p = 0.0011, Chi-squared — Responder Rate on Weekly CSBM1 in the ITT (Intention to Treat) analysis set. (For details, refer to the primary outcome description)
Statistical Analysis 2: Comparison: Vibrant Capsule Mode A vs Placebo Capsule; Test type: Superiority; p = 0.0085, Chi-squared — Responder Rate on Weekly CSBM2 in the ITT (Intention to Treat) analysis set. (For details, refer to the primary outcome description)

2. Secondary Outcome: Change From Baseline in Average Straining
Description: Change from baseline in average straining using (0-10) scale where "0" is no straining and "10" is unbearable straining
Time Frame: 8 weeks of treatment
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Vibrant Capsule Mode A | Placebo Capsule
Number analyzed (Participants) | 163 | 149
units on a scale | -1.56 [-1.90 to -1.22] | -1.0 [-1.40 to -0.60]

3. Secondary Outcome: Change From Baseline in Average Stool Consistency
Description: Change from baseline in average stool consistency, using the Bristol Stool Scale (1-7) where 1 = Separate hard lumps, like nuts (hard to pass) and 7 =watery, no solid pieces, entirely liquid
Time Frame: 8 weeks of treatment
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Vibrant Capsule Mode A | Placebo Capsule
Number analyzed (Participants) | 163 | 149
units on a scale | 0.92 [0.75 to 1.09] | 0.44 [0.24 to 0.64]

4. Secondary Outcome: Change From Baseline in Average Bloating
Description: Change from baseline in average bloating using scale (0-10) for bloating where 0=No bloating and 10=Unbearable bloating
Time Frame: 8 weeks of treatment
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Vibrant Capsule Mode A | Placebo Capsule
Number analyzed (Participants) | 163 | 149
units on a scale | -0.33 [-0.59 to -0.08] | -0.23 [-0.53 to 0.07]

5. Other Pre Specified Outcome: Change in SBM
Description: Change from baseline in weekly number of Spontaneous Bowel Movement (SBM)
Time Frame: 8 weeks of treatment
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: bowel movements/week
Arm/Group | Vibrant Capsule Mode A | Placebo Capsule
Number analyzed (Participants) | 163 | 149
bowel movements/week | 1.4 [1.08 to 1.73] | 1.24 [0.87 to 1.62]

6. Other Pre Specified Outcome: Change From Baseline in Quality of Life
Description: Change from baseline in average PAC-QOL (=Patient Assessment of Constipation Quality of Life) score.
  The results below present the number of participants who completed PAC-QOL questionnaire and reported an improvement in quality of life from baseline.
Time Frame: 8 weeks of treatment
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Vibrant Capsule Mode A | Placebo Capsule
Number analyzed (Participants) | 145 | 136
Participants | 113 | 90

ADVERSE EVENTS:
Time Frame: The Safety reporting conducted throughout the treatment period (8 weeks)
Groups:
- Vibrant Capsule Mode B: Vibrating capsule mode B administered 5 times per week. Based on the predefined interim analysis, mode B was discontinued, and the trial was completed using mode A. Therefore, only safety data was available for the dropped Arm B.
Arm/Group | Vibrant Capsule Mode A | Vibrant Capsule Mode B | Placebo Capsule
All-Cause Mortality (participants affected / at risk) | 0/163 | 0/37 | 0/149
Serious Adverse Events (participants affected / at risk) | 0/163 | 0/37 | 2/149
Other Adverse Events (participants affected / at risk) | 43/163 | 9/37 | 26/149
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vibrant Capsule Mode A (N=163) | Vibrant Capsule Mode B (N=37) | Placebo Capsule (N=149)
significant abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
transient ischemic attack (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Vibrant Capsule Mode A (N=163) | Vibrant Capsule Mode B (N=37) | Placebo Capsule (N=149)
Sensation of vibration (Product Issues) | 18 | 1 | 0 — Sensation of vibration was described as ''I think I felt vibration". Most patients did not find the sensation bothersome and none of the patients stopped the therapy due to this sensation.
Headache (Nervous system disorders) | 3 | 1 | 4
Urinary tract infection (Renal and urinary disorders) | 3 | 1 | 2
Abdominal pain (Gastrointestinal disorders) | 2 | 1 | 7
Abdominal discomfort (Gastrointestinal disorders) | 2 | 0 | 0
Vomiting (Gastrointestinal disorders) | 2 | 2 | 1
Nausea (Gastrointestinal disorders) | 3 | 0 | 1
Abdominal distention (Gastrointestinal disorders) | 1 | 0 | 2
Anorectal problem (Gastrointestinal disorders) | 1 | 0 | 4
Diarrhea (Gastrointestinal disorders) | 2 | 0 | 0
Covid-19 (Infections and infestations) | 1 | 0 | 2
Nasopharyngitis/ Bronchitis (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 3
Musculoskeletal (Musculoskeletal and connective tissue disorders) | 2 | 0 | 1
Fatigue (General disorders) | 2 | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Permission to use study data is required

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-01-24): https://cdn.clinicaltrials.gov/large-docs/39/NCT03879239/Prot_SAP_000.pdf